CLINICAL TRIAL: NCT01896492
Title: Clomiphene Citrate Plus N-acetyl Cysteine Versus Clomiphene Citrate for Induction of Ovulation in Women With Newly Diagnosed Polycystic Ovary Syndrome: a Randomized Double-blind Controlled Trial
Brief Title: Clomiphene Plus N-acetyl Cysteine for Induction of Ovulation in Newly Diagnosed Pcos.
Acronym: NACIPCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, alaa eldeen mahmoud ismail, M D, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: ccpnacinovi
Record Dates: First submitted 2013-06-22; First posted 2013-07-11 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: PCOS
Keywords: PCOS,; NAC,; OVULATION INDUCTION,; CLOMOPHEN CITRATE

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- N-acetyl cystien and clomiphen citrate (Active Comparator): N-acetyl cystien and clomiphen citrate,in induction of ovulation in newly diagnosed PCOS,1-2gm schats of NAC PLUS 100 mg of cc in the therd day of the cycle till day 8,with monitoring of follicular growth usin ultrasonography.HCG is giving to trigger of ovulation fo follicular size 18mm or more.
  Interventions: Drug: NAC
- Clomiphen citrate and placebo (Placebo Comparator): CC plus placebo compared to cc and NAC in induction of ovulation in PCOS new cases.
  Interventions: Drug: NAC
- N-acetyl cystien (No Intervention): In addition to the CC, each patient was selected randomly to receive either NAC (Sedico, Cairo, ARE), in a dose of 1.2 g/d orally, or a placebo (sugar) of the same volume twice daily from day 3 until day 7

INTERVENTIONS:
Drug: NAC — NAC 2gm plus cc 100mg from 3rd day of the cycle till day 8 with u/s follow up of the follicular growth.
  Other Names: N-acetyl cystien
  Arms: Clomiphen citrate and placebo; N-acetyl cystien and clomiphen citrate

SUMMARY:
Polycystic ovary syndrome (PCOS) is one of the most common endocrine disorders, affecting approximately 6-10% of women of reproductive age. Anovulation, infertility and hyperandrogenism often co-exist with hyperinsulinaemia and insulin resistance .

Clomiphene citrate remains the standard drug for induction or augmentation of ovulation. However, it is not equally effective in all situations, and therefore it may require additional expensive drugs such as N-acetyl cysteine, as an antioxidant, has been suggested as an adjuvant in clomiphene-resistant cases .NAC may also improve the circulating level of insulin and insulin sensitivity in hyperinsulinaemic women with PCOS, and may be useful for the treatment of insulin resistance by ameliorating the homocysteine and lipid profile in PCOS .

DETAILED DESCRIPTION:
NAC has been used effectively as an adjuvant to clomiphene citrate (CC) for ovulation induction in CC-resistant women with PCOS .

Because it is an insulin sensitizer, NAC was proposed as an adjuvant to clomiphene citrate for ovulation induction in patients with polycystic ovary syndrome who are resistant to clomiphene citrate. Encouraging results in those patients stimulated us to investigate whether adding NAC to the standard treatment with CC results in a higher ovulation rate, higher pregnancy rate, and less CC resistance in women with newly diagnosed polycystic ovary syndrome using a randomized, double-blind, controlled study.

ELIGIBILITY:
Inclusion Criteria:

* PCOS diagnosed by Rotterdam's criteria

Exclusion Criteria:

* previous induction of ovulation male factoe infertility tubal factor infertility uterine factor infertility

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Ovulation rate | 2 years
  Clomiphene citrate, 100 mg, was given from day 3 until day 7. In addition to the CC, each patient was selected randomly to receive either NAC (Sedico, Cairo, ARE), in a dose of 1.2 g/d orally, or a placebo (sugar) of the same volume twice daily from day 3 until day 7. Monitoring of the cycle will involve transvaginal determination of the mean follicular diameter and measurement of serum E2 levels. Monitoring intervals will be determined by patient response.

SECONDARY OUTCOMES:
include PR, number of follicles of ≥ 18 mm, the serum E2 concentration, serum P, and endometrial thickness | 2 years
  Clomiphene citrate, 100 mg, was given from day 3 until day 7. In addition to the CC, each patient was selected randomly to receive either NAC (Sedico, Cairo, ARE), in a dose of 1.2 g/d orally, or a placebo (sugar) of the same volume twice daily from day 3 until day 7. Monitoring of the cycle will involve transvaginal determination of the mean follicular diameter and measurement of serum E2 levels. Monitoring intervals will be determined by patient response. Human chorionic gonadotropin will be given when at least one follicle measured 18 mm and the E2 level had increased. Timed intercourse will be advised 24-36 hours after hCG injection. A serum P level will be checked on cycle days 21-22.
  A serum hCG level will be determined 14 days after hCG injection if menses had not yet occurred. Pregnancy will be defined as an increase in the serum hCG level on serial determinations at least 2 days apart.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Ismail, M D, Principal Investigator — Woman's Health University Hospital, Egypt